CLINICAL TRIAL: NCT02534597
Title: National Evaluation of Quality of Childcare (ENCCI)
Brief Title: National Evaluation of Quality of Childcare (C0682)
Acronym: ENCCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Whole Child International (Unknown); University of South Carolina (Other); University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jan Ostermann, Principal Investigator, Duke University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2017-0594
Record Dates: First submitted 2015-08-21; First posted 2015-08-27 (Estimated); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Child Rearing; Mental Health Wellness 1; Health Behavior
MeSH Terms: conditions — Health Behavior | interventions — Health Planning Technical Assistance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (10):
- pctm (Experimental): Receives the earliest Promotores training, followed by direct caregiver training, materials support, and technical assistance.
  Interventions: Behavioral: Promotores Training; Behavioral: Caregiver training; Behavioral: Materials support; Behavioral: Technical assistance
- p_ctm (Experimental): Receives the earliest Promotores training, followed by delayed caregiver training, delayed materials support, and delayed technical assistance.
  Interventions: Behavioral: Promotores Training; Behavioral: Delayed caregiver training; Behavioral: Delayed materials support; Behavioral: Delayed technical assistance
- _pmt (Experimental): Receives the delayed Promotores training, followed by receipt of materials support and technical assistance.
  Interventions: Behavioral: Delayed Promotores training; Behavioral: Materials support; Behavioral: Technical assistance
- _p_mt (Experimental): Receives the delayed Promotores training, followed by delayed receipt of materials support and technical assistance.
  Interventions: Behavioral: Delayed Promotores training; Behavioral: Delayed materials support; Behavioral: Delayed technical assistance
- _pct (Experimental): Receives the delayed Promotores training, followed by caregiver training and technical assistance.
  Interventions: Behavioral: Delayed Promotores training; Behavioral: Caregiver training; Behavioral: Technical assistance
- _p_ct (Experimental): Receives the delayed Promotores training, followed by delayed caregiver training and technical assistance.
  Interventions: Behavioral: Delayed Promotores training; Behavioral: Delayed caregiver training; Behavioral: Delayed technical assistance
- _pt (Experimental): Receives the delayed Promotores training, followed by technical assistance.
  Interventions: Behavioral: Delayed Promotores training; Behavioral: Technical assistance
- _p_t (Experimental): Receives the delayed Promotores training, followed by delayed technical assistance.
  Interventions: Behavioral: Delayed Promotores training; Behavioral: Delayed technical assistance
- _pc (Experimental): Receives the delayed Promotores training, followed by a full caregiver training only.
  Interventions: Behavioral: Delayed Promotores training; Behavioral: Caregiver training
- _p_c (Experimental): Receives the delayed Promotores training, followed by delayed caregiver training.
  Interventions: Behavioral: Delayed Promotores training; Behavioral: Delayed caregiver training

INTERVENTIONS:
Behavioral: Promotores Training
  Arms: p_ctm; pctm
Behavioral: Delayed Promotores training
  Arms: _p_c; _p_ct; _p_mt; _p_t; _pc; _pct; _pmt; _pt
Behavioral: Caregiver training
  Arms: _pc; _pct; pctm
Behavioral: Delayed caregiver training
  Arms: _p_c; _p_ct; p_ctm
Behavioral: Materials support
  Arms: _pmt; pctm
Behavioral: Delayed materials support
  Arms: _p_mt; p_ctm
Behavioral: Technical assistance
  Arms: _pct; _pmt; _pt; pctm
Behavioral: Delayed technical assistance
  Arms: _p_ct; _p_mt; _p_t; p_ctm

SUMMARY:
This evaluation seeks to assess the impact of a training program on childcare center environments and child/caregiver wellbeing in El Salvador. Through a longitudinal, randomized control trial, over 200 childcare centers participating in the program will be assigned to various treatment arms receiving different components of the program. A community comparison cohort will also be enrolled.

DETAILED DESCRIPTION:
Whole Child International (WCI) is a U.S.-based non-governmental organization. Its focus is on improving the caregiving environments for vulnerable children by effecting changes within child care centers and orphanages.

This evaluation will assess the impact of an educational training and technical assistance program offered by WCI in collaboration with the El Salvadoran government. The program consists of a series of educational trainings (for local government officials, directors of childcare and residential centers, and center caregivers) and technical assistance including infrastructural changes within centers.

To evaluate this intervention, a longitudinal, randomized controlled trial will be used to assign participating centers to one of seven treatment arms that will receive different components of the intervention. A community comparison cohort will also be enrolled to identify selection effects as well as local norms and standards. The central research question is, "Does providing training for institution providers and caregivers improve child outcomes?"

Ethnographic research will also explore local cultural norms regarding child caregiving, and seek to understand how the intervention is received within communities.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 6 months-4 years old at baseline, who are currently attending government-run childcare centers in El Salvador, will be eligible for enrollment in this study. One parent/guardian and center caregiver for an enrolled child will also complete assessments.
* In the comparison group, for every 5th center-attending child enrolled, the nearest neighboring child between the ages of 6 months and 4 years at enrollment, and who does not attend the center, will be eligible for enrollment. One parent/guardian of the comparison child will also complete assessments.

Exclusion Criteria:

* Children with known disabilities, who are unlikely to show developmental changes over time, may be excluded from the study.

Ages: 6 Months to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1923 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Children's developmental milestone achievement as measured by the Battelle Developmental Inventory, Second Edition (BDI-2). | Four years
  The BDI-2 Developmental Quotient has a mean of 100, standard deviation of 15, score range 40-160.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Ostermann, PhD, Principal Investigator — Associate Research Professor; Kathryn Whetten, PhD, Principal Investigator — Professor
Locations (1):
- Whole Child International, San Salvador, El Salvador